CLINICAL TRIAL: NCT03847792
Title: Analgesic Effect Of Intra-articular Dexamethasone Versus Fentanyl Added as an Adjuvant to Bupivacaine for Postoperative Pain Relief in Knee Arthroscopic Surgery
Brief Title: Analgesic Effect Of Intra-articular Bupivacaine Fentanyl for Postoperative Pain Relief in Knee Arthroscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MS/18.09.306
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Knee Arthroscopic Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group DB/Dexamethasone-Bupivacaine (Active Comparator): Patients were received an intra-articular injection of 8mg dexamethasone added to18mL of 0.25% bupivacaine
  Interventions: Drug: Group DB/Dexamethasone-Bupivacaine
- Group FB /Fentanyl-Bupivacaine (Active Comparator): Patients were received an intra-articular injection of 1 ug/kg fentanyl added to 18 mL of 0.25% bupivacaine
  Interventions: Drug: Group FB /Fentanyl-Bupivacaine
- Group PB/Placebo-Bupivacaine (Placebo Comparator): Patients were received an intra-articular injection of 2 mL isotonic saline added to 18 mL of 0.25% bupivacaine
  Interventions: Drug: Group PB/Placebo-Bupivacaine

INTERVENTIONS:
Drug: Group DB/Dexamethasone-Bupivacaine — The patient were received an intra-articular injection of 18ml bupivacaine 0.25% added to 8mg dexamethasone.
  Arms: Group DB/Dexamethasone-Bupivacaine
Drug: Group FB /Fentanyl-Bupivacaine — The patient were received an intra-articular injection of 1 ug/kg fentanyl added to 18ml of 0.25% bupivacaine.
  Arms: Group FB /Fentanyl-Bupivacaine
Drug: Group PB/Placebo-Bupivacaine — Patients were received an intra-articular injection of 2ml isotonic saline added to 18ml of 0.25% bupivacaine.
  Arms: Group PB/Placebo-Bupivacaine

SUMMARY:
However, local anesthetic agents can produce analgesia for a limited time when used as a single injection. Bupivacaine is a local anesthetic that has an immediate action on pain by blocking peripheral afferents. However, as the ideal analgesic, the drug must cover the whole postoperative period (≥ 24 hours); therefore, bupivacaine is usually combined with many adjutants to provide long-lasting post-arthroscopy analgesia.

DETAILED DESCRIPTION:
Intr-articular drug administration has gained popularity because of its simplicity and efficacy in achieving anesthesia for diagnostic and operative arthroscopy and for providing postoperative analgesia .although the knee joint has been examined most commonly, arthroscopy of other joints such as shoulder, ankle, wrist, metatarsophalangeal and temporomandibular joints is being increasingly used.

Intra-articular installation of local anesthesia during arthroscopic procedures has been used by many orthopedic surgeons to provide pain relief after surgery.The aim of this study was to evaluate the analgesic efficacy of intra-articular dexamethasone versus fentanyl added as an adjuvant to bupivacaine in patients undergoing knee arthroscopic surgery

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status (ASA) I or II

Exclusion Criteria:

* Contraindication to spinal anesthesia.
* Allergy to the study drugs.
* Refusal of the patients.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2019-03-31 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | for 24 hour after surgery
  Time to the first request of pethidine in minutes within the first 24 hours postoperatively

SECONDARY OUTCOMES:
Total analgesic requirement | for 24 hour after surgery
  Total analgesic requirement of pethidine will be recorded during the first 24 hours following surgery
Mean arterial blood pressure | At 1,2,4,6,8,12,18 and 24 hours postoperatively.
  Mean arterial blood pressure measured in mm Hg and assessed at 1,2,4,6,8,12,18 and 24 hours following the discharge of the patient from the operating theatre.
Heart rate | At 1,2,4,6,8,12,18 and 24 hours postoperatively.
  Heart rate will be measured in beats/minute and assessed at 1,2,4,6,8,12,18 and 24 hours following the discharge of the patient from the operating theatre.
Pain score | measured at 1,2,4,6,8,12,18 and 24 hours postoperatively.
  Measured with visual analogue score(VAS):0=no pain and 100=worst imaginable pain measured at 1,2,4,6,8,12,18 and 24 hours
Patients' satisfaction | for 24 hour after surgery
  satisfaction score from 1 to 4; as 4=Excellent ,3=good ,2=satisfactory and 1=poor will be measured after 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Sultan, MD, Study Chair — Professor of Anaesthesia and Surgical Intensive Care; Hazem ESM Weheba, MD, Study Director — Assistant Professor of Anaesthesia and Surgical Intensive Care; Hosam Ibrahim EL said saber, MD, Study Director — Lecturer of Anaesthesia and Surgical Intensive Care
Locations (2):
- Egypt (2):
  - Mohamed A Sultan, Al Mansurah, DK
  - Mansoura University, Al Mansurah, Eastern

IPD SHARING:
Plan to Share IPD: Yes
Following publication
Supporting Information: Study Protocol
Time Frame: forever
Access Criteria: tawfik20192@gmail.com